**Title:** Prophylactic antibiotic use in transarterial chemoembolization for hepatocellular carcinoma: an open-label, randomised, prospective study

#### **Introduction:**

Liver cancer especially hepatocellular carcinoma (HCC) is among the top five most common carcinomas in the world [1]. The treatment options for HCC includes surgery, liver transplantation, and radiofrequency ablation (RFA) with good survival rates. However, most HCC patients have angioinvasion. Furthermore, multiple lesions cannot be treated with such treatment strategies [2]. Image-guided transarterial chemoembolization (TACE) is accepted worldwide as a standard of care treatment for patients with hepatocellular carcinoma (HCC) in intermediate stage and good performance status [3]. TACE procedures, performed by the interventional radiologists, are minimally invasive with excellent outcomes as part of the nonsurgical treatment of HCC [1, 4]. Post-procedure-infection is uncommon but can lead to liver abscess and prolonged hospital stay. [7, 8] The chances of post-procedure-infection are higher in patients taking anticancer drugs due to immunosupression. [5, 6]. Incidence of liver abscess after TACE is 0.1 - 4.5% but carries a mortality rate of up to 50% [7, 8, 9].

TACE was linked to a risk of liver abscess. Prophylactic antibiotics pre-procedure lower this risk and ensuing surgical intervention [6]. Prophylactic antibiotics may not be required in TACE for HCC patients [10, 11, 12]. Moreover, old age, compromised hepatic function, hypoalbuminemia, portal vein cancer embolus, invasive procedures, using broad-spectrum antibiotics, and having diabetes mellitus are the independent risk factors for hospital-acquired infections (HAIs) after TACE in patients with primary liver cancer [1, 13].

According to the latest Cardiovascular and Interventional Radiological Society of Europe (CIRSE) standards of practice guidelines (2021), routine antibiotic prophylaxis is not recommended [14]. However, prophylactic antibiotics are recommended in cases where there is a high risk of developing a liver abscess. These include biliary obstruction or the presence of a bilioenteric anastomosis. The choice of agent is dependent on the suspected path ogens (upper gastrointestinal tract flora) and consideration should be given to potential hepatotoxicity of each agent. In complex cases involving multiple organisms, antibiotic resistance, or allergies, consulting with a microbiologist may be beneficial [14].

To date, it is uncertain whether the use of antibiotics as prophylaxis before TACE is beneficial or not in the prevention of postoperative infection.

Excessive antibiotic use is a global problem and carries risks of adverse drug reactions like allergy or anaphylaxis, increased cost, and contributes to the emergence antimicrobial resistance [15, 16]. Therefore, it is the need of the hour to explore the utility of prophylactic antibiotics in TACE.

This study aims to determine the effectiveness of prophylactic antibiotic use for TACE and occurrence of postoperative liver abscess.

## Methods

#### **Inclusion Criteria:**

- 1. Age 18 65 years
- 2. Diagnosis of primary liver cancer or hepatocellular carcinoma
- 3. Patients receiving TACE in PKLI & RC

## **Exclusion Criteria:**

- 1. Receiving two or more TACE during the same hospitalization
- 2. Use of any antibiotics other than the prophylactic antibiotic in 48hours prior to TACE
- 3. Known hypersensitivity to specified antibiotic used in the study
- 4. Incomplete or missing laboratory investigations and data
- 5. Taking Sorafenib before TACE
- 6. TACE combined with ablation or immunetherapy
- 7. Tumor size >10 cm
- 8. Portal vein thrombosis
- 9. Dilated biliary channels on CT scan / Billiary invasion by tumor

# **Study Outcomes:**

- 1. Predominantly neutrophilic leukocytosis (  $> 11 \times 10^9$ /L) with fever ( > 38 °C) in upto 48 hours post-TACE
- 2. Occurrence of liver abscess as diagnosed by imaging within 30 days of the procedure

3. Liver abscess requiring an intervention (e.g., percutaneous transhepatic abscess drainage (PTAD), percutaneous transhepatic abscess puncture or liver abscess incision) within 30 days of TACE

# **Sampling Technique:**

In this study, consecutive sampling technique and randomization by lottery method will be applied. In lottery method the investigator will randomly draw numbers from the box to choose sample until the final sample size reaches. Two numbers will be assigned as '1' for antibiotic group and '2' for no antibiotic group.

Current standard of care treatment at PKLI&RC (as per local guidelines) would be given to all patients receiving TACE for the intervention group or 'antibiotic group' (i.e., Inj. Ceftriaxone 1g, intravenous × stat). While no antibiotic would be given to the 'no antibiotic group'.

# Statistical analysis:

- 1. Data to be recorded on Excel sheet and subsequently exported to SPSS version 24 for further analysis.
- 2. A univariate analysis will be employed for the comparison of variations in patients' baseline characteristics between the preventive medication group and the nonpreventive medication group. The Student's t-test will be employed to evaluate if the obtained data had a homogeneous variance and a normal distribution. For nonhomogeneous variance, the comparisons were made using a one-way analysis of variance (ANOVA). In order to compare categorical variables, Fisher's exact test or Pearson's 2 test was used as applicable.
- 3. The univariate analysis included chi-square tests for categorical variables and t-tests for continuous variables. Significant variables (P < 0.01) in univariate analysis and covariates considered clinically influential were then analyzed by multivariate stepwise logistic regression (forward stepwise logistic regression) to identify significant variables. We applied univariate and multivariate logistic regression models to estimate odds ratios (ORs) with 95% confidence intervals (CIs) for significant

- variables for finding potential risk factors in WBC> $11\times10^9$ /L group or postoperative infection group.
- 4. *P* value less than 0.05 was considered statistically significant.

## **References:**

- Li B. Prophylactic Use of Antibiotics for Postsurgical Infection in c-TACE and DEB-TACE High-Risk Patients: A Case-Control Study. Journal of Healthcare Engineering. 2022 Apr 11;2022.
- 2. Chan WH, Huang SF, Lee CW, Wu TH, Pan KT, Lin SM, Yu MC, Hung CF. Incorporation of biochemical factors for survival analysis of transarterial chemoembolization in patients with hepatocellular carcinoma: A retrospective cohort study. Journal of International Medical Research. 2019 Oct;47(10):4862-71.
- 3. Mansour MA, Khalifa MO. Antibiotic prophylaxis in transarterial chemoembolization of hepatocellular carcinoma. Arab journal of gastroenterology. 2018 Mar 1;19(1):16-20.
- 4. Kang SJ, Kim UJ, Kim SE, An JH, Jang MO, Myung DS, Park KH, Jung SI, Cho SB, Jang HC, Joo YE. Predictive value of procalcitonin for bacterial infection after transarterial chemoembolization or radiofrequency ablation for hepatocellular carcinoma. Disease Markers. 2018 Apr 17;2018.
- 5. Dutta R, Mahato RI. Recent advances in hepatocellular carcinoma therapy. Pharmacology & therapeutics. 2017 May 1;173:106-17.
- 6. Yoshihara S, Yamana H, Akahane M, Kishimoto M, Nishioka Y, Noda T, Matsui H, Fushimi K, Yasunaga H, Kasahara K, Imamura T. Association between prophylactic antibiotic use for transarterial chemoembolization and occurrence of liver abscess: a retrospective cohort study. Clinical Microbiology and Infection. 2021 Oct 1;27(10):1514-e5.
- 7. Song SY, Chung JW, Han JK, Lim HG, Koh YH, Park JH, Lee HS,Kim CY. Liver abscess after transcatheter oily chemoembolization for hepatic tumors: incidence, predisposing factors, and clinical outcome. J Vasc Interv Radiol. 2001;12(3):313–20.
- 8. Yang C, Tsauo J, Li X. Liver abscess after transcatheter arterial chemoembolization for hepatocellular carcinoma: clinical manifestations, risk factors, diagnosis, prevention, and treatment. Chinese Journal of Academic Radiology. 2022 Mar 12:1-5.

- 9. Shin JU, Kim KM, Shin SW, Min SY, Park SU, Sinn DH, Gwak GY, Choi MS, Lee JH, Paik SW, Yoo BC. A prediction model for liver abscess developing after transarterial chemoembolization in patients with hepatocellular carcinoma. Digestive and Liver Disease. 2014 Sep 1;46(9):813-7.
- 10. Shi Z, Yang W, Tang H, Li X. Risk factors of infection after transarterial chemoembolization for hepatocellular carcinoma: a protocol for systematic review and meta-analysis. Medicine. 2021 May 5;100(20).
- 11. Plentz RR, Lankisch TO, Bastürk M, Müller CC, Kirchhoff T, Gebel M, Bleck JS, Kubicka S, Manns MP, Meier PN, Rudolph KL. Prospective analysis of German patients with hepatocellular carcinoma undergoing transcatheter arterial chemoembolization with or without prophylactic antibiotic therapy. Journal of gastroenterology and hepatology. 2005 Jul;20(7):1134-6.
- 12. Castells A, Bruix J, Ayuso C, Brú C, Montayà X, Boix L, Rodès J. Transarterial embolization for hepatocellular carcinoma. Antibiotic prophylaxis and clinical meaning of postembolization fever. Journal of hepatology. 1995 Apr 1;22(4):410-5.
- 13. Nouri YM, Kim JH, Yoon HK, Ko HK, Shin JH, Gwon DI. Update on transarterial chemoembolization with drug-eluting microspheres for hepatocellular carcinoma. Korean Journal of Radiology. 2019 Jan 1;20(1):34-49.
- 14. Lucatelli P, Burrel M, Guiu B, de Rubeis G, van Delden O, Helmberger T. CIRSE standards of practice on hepatic transarterial chemoembolisation. Cardiovascular and Interventional Radiology. 2021 Dec;44(12):1851-67.
- 15. Costelloe C, Metcalfe C, Lovering A, Mant D, Hay AD. Effect of antibiotic prescribing in primary care on antimicrobial resistance in individual patients: systematic review and meta-analysis. Bmj. 2010 May 18;340.
- 16. Nepal G, Bhatta S. Self-medication with antibiotics in WHO Southeast Asian Region: a systematic review. Cureus. 2018 Apr 5;10(4).